CLINICAL TRIAL: NCT02946216
Title: Frequency and Abundance of ALK/ROS1/MET Mutations on Circulating Tumor DNA in Patients With Non-small Cell Lung Cancer Using Single Molecule Amplifcation and Re-sequencing Technology: a Perspective Observational Study
Brief Title: ALK/ROS1/MET Mutations on Plasma ctDNA in Patients With NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-101-01
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Non-small Cell Lung Cancer Stage III; Non-Small-Cell Lung Cancer Metastatic; Adenocarcinoma of Lung; EGFR Wildtype
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: ctDNA analysis

SUMMARY:
The study aims to explore the prevalence of ALK/ROS1/MET mutations assessed with ctDNA samples in EGFR-wildtype NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB/IV NSCLC;
* Histologically confirmed adenocarcinoma;
* EGFR-wildtype NSCLC;
* Provision of blood (plasma) sample for ctDNA testing;
* Patient must be able to comply with the protocol;
* Provision of blood (plasma) sample for ctDNA testing;

Exclusion Criteria:

* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease);
* Histologically confirmed small cell lung cancer or other metastatic tumors;
* Patient with no histologic or cytological diagnosis;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ALK/ROS1/MET mutations detected by single molecule amplifcation and re-sequencing technology (cSMART) | up to 2 years
  The investigators will describe the proportion of ALK/ROS1/MET mutations on ctDNA detected by cSMART in patients with non-small cell lung cancer (NSCLC)
Proportion of patients with ALK/ROS1/MET mutations detected by single molecule amplifcation and re-sequencing technology (cSMART) after crizotinib resistance | up to 2 years
  The investigators will describe the proportion of ALK/ROS1/MET mutations on ctDNA detected by cSMART in patients with non-small cell lung cancer (NSCLC) after crizotinib resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Nanjing Medical University, Hangzhou, Zhejiang, China